CLINICAL TRIAL: NCT02702154
Title: A Randomized Sham-Controlled Study of High- and Low-frequency Repetitive Transcranial Magnetic Stimulation of the Dorsomedial Prefrontal Cortex in Major Depressive Disorder
Brief Title: High-frequency vs. Low-frequency vs. Sham DMPFC-rTMS for Major Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jonathan Downar, Co-Director, UHN MRI-Guided rTMS Clinic, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-9276-A
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: brain stimulation; rTMS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-frequency rTMS (Experimental): 20 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, twice daily, 5 days per week for 3 weeks
  Interventions: Device: High-frequency rTMS
- Low-frequency rTMS (Experimental): 1 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, twice daily, 5 days per week for 3 weeks
  Interventions: Device: Low-frequency rTMS
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, twice daily, 5 days per week for 3 weeks
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: High-frequency rTMS — 20 Hz active stimulation, twice daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: High-frequency rTMS
Device: Low-frequency rTMS — 1 Hz active stimulation, twice daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: Low-frequency rTMS
Device: Sham rTMS — Sham stimulation, twice daily
  Other Names: Magventure Cool DB80 Active/Placebo Coil
  Arms: Sham rTMS

SUMMARY:
This trial will compare the efficacy and tolerability of 20 Hz vs. 1 Hz vs. sham repetitive transcranial magnetic stimulation targeting the dorsomedial prefrontal cortex, delivered twice daily over 15 days, in patients with a diagnosis of major depressive disorder. The trial will include structural and functional MRI, EEG, and behavioral measures obtained before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria (Patient):

* Voluntary and competent to consent to treatment
* MINI confirmed diagnosis of MDD
* Outpatient
* Between the ages of 18-65
* Failed to achieve a clinical response to at least one pharmacotherapy or behavioral treatment in the current episode.
* Have had no increase or initiation of any psychotropic medication in the last 4 weeks prior to screening
* Must adhere to study assessment and intervention schedule.
* Pass the TMS Safety Screening Questionnaire.

Exclusion Criteria (Patient):

* Have a concomitant major unstable medical illness, cardiac pacemaker or implanted medical pump
* Have active suicidal intent
* Are pregnant
* Have a lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms have a MINI diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia assessed by a study investigator to be primary and causing greater impairment than MDD
* Have received rTMS for any previous indication due to the potential compromise of subject blinding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
HAM-D17 score | Baseline, after each week (10 sessions) of treatment, and 2, 6, and 12 weeks post-treatment
  Outcome measured by a change in HAM-D17 score from baseline to 2 weeks post-treatment. A 50% improvement in the score is considered a response to rTMS. A final score of <8 is categorized as remission.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | Baseline, after each week (10 sessions) of treatment, and 2, 6, and 12 weeks post-treatment
Beck anxiety inventory | Baseline, after each week (10 sessions) of treatment, and 2, 6, and 12 weeks post-treatment

OTHER OUTCOMES:
Resting-state functional MRI | 1 week pre- and 1 week post-intervention
  10 min resting-state functional MRI acquisition at 3T
Electroencephalography | Day 1 and day 15 (final day) of rTMS intervention
  10 min resting-state and task-based (response inhibition, reward sensitivity) acquisitions

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Downar, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided